CLINICAL TRIAL: NCT04208516
Title: A Prospective, Randomized, Active-Comparator, Open-Label, Non-Inferiority Study of the Efficacy of Continuous Nerve Block vs Single Block Plus Intravenous Lidocaine for Postoperative Pain.
Brief Title: Continuous Nerve Block Block vs Combination of Single Block Plus Intravenous Lidocaine for Postoperative Pain.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was unable to be obtained in a timely fashion, so the study was stopped.
Sponsor: Jeremy Kearns (Other)
Responsible Party: Sponsor-Investigator, Jeremy Kearns, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19100057
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
Keywords: intravenous lidocaine; erector spinae plane block; quadratus lumborum block; thoracic surgery; abdominal surgery; continuous peripheral nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexamethasone; Dexmedetomidine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Two groups of patients will be studied simultaneously. One group will receive continuous peripheral nerve blocks and the other group will receive single blocks plus postoperative intravenous lidocaine infusion.
Who Masked: Outcomes Assessor
Masking Description: For study participants, the investigator placing the block will record in the narrative that "this patient is a study participant and received Paravertebral block with ESP approach" or "this patient is a study participant and received TAP block with QL approach". By documenting blocks in this way, the research team member collecting the data will be blinded to whether the patient received continuous block with 0.5% ropivacaine, or single block with 0.5% ropivacaine, dexamethasone, and dexmedetomidine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous nerve blocks (Active Comparator): A total of 30 subjects equally distributed to either continuous Erector Spinae Plane block for unilateral thoracic surgery , or continuous Quadratus Lumborum block for major abdominal surgery. Patients in this group will receive 20ml 0.5% ropivacaine per block performed after positioning of the needle followed by continuous perineural infusion of 0.25% lidocaine (10ml/hr) beginning in the post-anesthesia care unit (PACU) and continued for 72 hours or until 12 hours prior to patient discharge, whichever comes first, which is standard of care at this institution.
  Interventions: Procedure: Continuous Erector Spinae Plane Nerve Block; Procedure: Continuous Quadratus Lumborum Nerve Block; Drug: Ropivacaine 0.5% Injectable Solution; Drug: Lidocaine
- Single nerve blocks plus IV lidocaine infusion (Experimental): A total of 30 subjects equally distributed to either Erector Spinae Plane block for unilateral thoracic surgery, or Quadratus Lumborum block for major abdominal surgery, will be included . Patients in this group will receive 20ml 0.5% ropivacaine, 4mg dexamethasone, and 20mcg dexmedetomidine (30mcg if only one block is performed) per block after proper positioning of the Tuohy needle. Upon patient arrival in the recovery room a continuous infusion of IV lidocaine 50 mg /hr will be started and continued for 72 hours or until 12 hours prior to patient discharge, whichever comes first, which is standard of care at this institution.
  Interventions: Procedure: Single Erector Spinae Plane Nerve Block; Procedure: Single Quadratus Lumborum Nerve Block; Drug: Lidocaine IV; Drug: Ropivacaine 0.5% Injectable Solution; Drug: Dexamethasone; Drug: Dexmedetomidine

INTERVENTIONS:
Procedure: Continuous Erector Spinae Plane Nerve Block — To be administered to subjects in the active comparator group receiving primary unilateral thoracic surgery.
  Arms: Continuous nerve blocks
Procedure: Continuous Quadratus Lumborum Nerve Block — To be administered to subjects in the active comparator group receiving primary major abdominal surgery.
  Arms: Continuous nerve blocks
Procedure: Single Erector Spinae Plane Nerve Block — To be administered to subjects in the experimental group receiving primary unilateral thoracic surgery.
  Arms: Single nerve blocks plus IV lidocaine infusion
Procedure: Single Quadratus Lumborum Nerve Block — To be administered to subjects in the experimental group receiving primary major abdominal surgery.
  Arms: Single nerve blocks plus IV lidocaine infusion
Drug: Lidocaine IV — To be given postoperatively as a continuous infusion at a dose of 50 mg/hr in the experimental group.
  Arms: Single nerve blocks plus IV lidocaine infusion
Drug: Ropivacaine 0.5% Injectable Solution — To be used in both treatment arms as nerve block initial bolus injection.
Drug: Dexamethasone — To be used in the experimental arm as a nerve block adjuvant to promote prolonged single block duration, as is standard of care in this institution.
  Arms: Single nerve blocks plus IV lidocaine infusion
Drug: Dexmedetomidine — To be used in the experimental arm as a nerve block adjuvant to promote prolonged single block duration, as is standard of care in this institution.
  Arms: Single nerve blocks plus IV lidocaine infusion
Drug: Lidocaine — To be used perineurally as a 0.25% solution in the active comparator group at a rate of 10 ml/hr per perineural catheter.
  Arms: Continuous nerve blocks

SUMMARY:
A multimodal analgesic regimen including regional anesthesia is used at UPMC Shadyside for primary thoracic and major abdominal surgeries. The current standard-of-care regional anesthesia techniques include Erector Spinae Plane (ESP) block for video assisted thorascopic surgery (VATS) and Quadratus Lumborum (QL) block for major abdominal surgery. These blocks are routinely administered as a continuous catheter technique in order to extend the duration of postoperative analgesia. Although rare, continuous nerve block techniques carry risks and limitations, including catheter dislodgement, migration, kinking and leaking at the site, bleeding, and infection. They are also much more expensive to perform and maintain than single-injection nerve blocks at this institution. Perioperative intravenous (IV) lidocaine is one of the safest local anesthetics, and its use has been shown to provide analgesia and reduce opioid requirements. Furthermore, it has been hypothesized that part of the analgesic efficacy of continuous peripheral nerve blocks may be due to the systemic effects of the local anesthetic infused at the site. Therefore, it is possible that the combination of a single block followed by an infusion of IV lidocaine may provide the same benefits as a continuous nerve block at a lower cost. The purpose of this study is to show that a single block technique plus IV lidocaine is non-inferior to a continuous block technique. For the purpose of this study we chose two surgical models--VATS and major abdominal surgery--and ESP and QL blocks, respectively. The study will be conducted as a prospective, randomized (1:1), open-label, active-comparator, noninferiority trial. The study will prospectively investigate the efficacy of continuous block versus single block plus IV lidocaine infusion for postoperative pain management in patients undergoing primary unilateral VATS or primary major abdominal surgery.

DETAILED DESCRIPTION:
After obtaining a signed informed consent, participating patients will be randomized by computer generated random numbers to either the control group to receive continuous Erector Spinae Plane block (in the case of thoracic surgery) or continuous Quadratus Lumborum block (in the case of abdominal surgery), or the treatment group to receive single shot Erector Spinae Plane block (in the case of thoracic surgery) or single shot Quadratus Lumborum block (in the case of abdominal surgery) with postoperative intravenous lidocaine infusion. Subjects will be randomized in a 1:1 ratio. Randomization will take place via an opaque envelope containing the treatment group allocation that will be given to the anesthesiologist performing the block after informed consent is signed. Procedures will take place in the UPMC Shadyside pre-operative block area. The expected duration of nerve block procedures is 10-20 minutes.

If the patient is randomized to the continuous nerve block group and is undergoing thoracic surgery, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach:

Continuous ESP Block Approach: The patient will be positioned in seated position with side or sides to be blocked marked. The T5 spinous process will be identified by palpation starting with C7 and continuing caudad. C7 is the most prominent spinous process anatomically. The T5 spinous process will be marked with a marking pen. The block area will be cleaned using 2% chlorhexidine solution. The entire block procedure is performed under strict aseptic technique. An ultrasound probe covered in a sterile probe cover will be placed at the T5 spinous process in a cephalad to caudad orientation and moved lateral until the T5 transverse process is identified. 1-2ml of 1% lidocaine will be administered just above the ultrasound probe for local skin infiltration. An 18 gauge Tuohy needle will then be inserted in plane in a cephalad to caudad direction under ultrasound visualization until the tip of the needle touches the T5 transverse process. The T5 transverse process is the anatomical target for this block. 20ml of 0.5% ropivacaine will then be injected using slow fractionated injection, aspirating every 5ml to ensure the needle tip is not intravascular. Local anesthetic spread in the appropriate plane will be confirmed with ultrasound. Once injection is complete, a 20 gauge nonstimulating catheter will be inserted through the Tuohy needle. Catheter tip placement will be confirmed with ultrasound. If bilateral blocks are to be performed, the procedure will then be repeated on the contralateral side. Upon patient arrival to PACU, a continuous infusion of 0.25% lidocaine at 10ml/hr per side blocked via ESP catheter will be initiated and continued for 72 hours or until 12 hours prior to patient discharge.

If the patient is randomized to the continuous nerve block group and is undergoing abdominal surgery, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach:

Continuous QL Block Approach: The patient will be positioned in lateral decubitus position with the side to be blocked facing up and the side or sides to be blocked marked. The block area will be cleaned using 2% chlorhexidine solution. The entire block procedure is performed under strict aseptic technique. An ultrasound probe covered in a sterile probe cover will be placed transversally between the iliac crest and the costal margin at the level of the anterior axillary line and the three muscles of the anterolateral abdominal wall (external oblique, internal oblique and transversus abdominis) will be identified. The probe will then be moved posteriorly until the transversus abdominis muscle (TAM) tapers off into its aponeurosis approximately at the level of the posterior axillary line, and posteriorly to this the intersection of the transversalis fascia with the lateral side of the QL muscle will be identified. An 18 gauge Tuohy needle will then be inserted in plane in an anterior to posterior direction until the tip of the needle is visualized at the intersection of the transversalis fascia with the lateral side of the QL muscle. The intersection of the transversalis fascia with the lateral side of the QL muscle is the anatomical target for this block. Once the initial injection of local anesthetic is complete, a 20 gauge nonstimulating catheter will be inserted through the Tuohy needle. Catheter tip placement will be confirmed with ultrasound. If bilateral blocks are to be performed, the patient will be repositioned, the area to be blocked will be cleaned and prepared in a strict aseptic fashion as described above, and the procedure will then be repeated on the contralateral side. Upon patient arrival to PACU, a continuous infusion of 0.25% Lidocaine at 10ml/hr per side blocked via QLB catheter will be initiated and continued for 72 hours or until 12 hours prior to patient discharge.

If the patient is randomized to the single block plus IV lidocaine group and is undergoing thoracic surgery, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach:

Single Shot ESP Block with Postoperative IV Lidocaine Approach: The same technique described for the CESP will be used except that in this case a single ESP block will be performed. A 22 gauge Tuohy needle will be used to perform these blocks. After the proper positioning of the needle 20ml of 0.5% ropivacaine plus, 4mg dexamethasone, plus 30mcg dexmedetomidine will be deposited. In the recovery room an infusion of IV lidocaine at 50mg/hr for be initiated for 72 hours or until 12 hours prior to patient discharge.

If the patient is randomized to the single block plus IV lidocaine group and is undergoing abdominal surgery, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach:

Single Shot QL Block with Postoperative IV Lidocaine Approach: The same technique described for the CQL will be used except that a single QL block will be performed. A 22 gauge Tuohy needle will be used to perform these blocks. After the proper positioning of the needle 20ml of 0.5% ropivacaine plus, 4mg dexamethasone, plus 20mcg dexmedetomidine per injection site (30mcg if unilateral block only) will be deposited. Upon patient arrival to PACU, a continuous infusion of intravenous lidocaine at 50mg/hr will be initiated and continued for 72 hours or until 12 hours prior to patient discharge.

Anesthetic Management: Both treatment groups will receive the standard anesthetic technique and multimodal analgesic technique at our institution, including preoperative gabapentin 300mg PO and acetaminophen 1000mg PO, intraoperative IV propofol infusion-based general anesthetic combined with sub-anesthetic dose IV ketamine infusion, IV dexmedetomidine infusion, IV acetaminophen, and avoidance of intraoperative opioids. Postoperative pain management will also follow standard protocol, using IV hydromorphone (0.2-0.3 mg) and PO oxycodone (5-10 mg) on request by the patient for moderate to severe pain (VAS >5), scheduled ketamine 20-50mg PO q 8hrs for 48 hours, scheduled acetaminophen 1000mg IV or PO q 6hrs, scheduled gabapentin 100-300mg PO at bedtime, and dexmedetomidine infusion 0.2mcg/kg/hr IV for 24 hours if the patient is located in the Intensive Care Unit.

After surgery, the patient will be followed by the blinded research team for incidence of adverse events, as well as the collection of the primary and secondary outcome measures. Pain assessment will be done by nurses in the PACU and on the floor using Numeric Pain Rating Scale, with 0 meaning no pain and 10 meaning worst possible pain. Opioid medication consumption, pain scores, local anesthetic medication consumption, serum lidocaine levels, and adverse effects will be recorded on worksheets included in patient research folders, with each study participant having their own research folder identified only by randomly assigned patient study number.

The research coordinator responsible for data collection will remain blinded to the patient's group allocation, and will not become unblinded during the data collection process because data will be collected from the patient's medical record and will not involve physically observing the patient (which would otherwise result in unblinding since the presence or absence of a perineural catheter and patient pump status would make the group allocation obvious). However, this information will not be obtainable when collecting data from the medical record. It is not possible to blind nursing staff or the patient to the patient's group allocation because the presence or absence of a visible perineural catheter will make the group allocation obvious.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* Primary unilateral VATS or major abdominal surgery
* BMI 20-36, weight ≥ 50kg
* Male and Female
* All races

Exclusion Criteria:

* Patient refusal
* Inpatient status at the time of surgery
* ASA class 4 or greater
* Pregnancy
* Non-English speaking or inability to participate in the study
* Patients with coagulopathy or on therapeutic anticoagulation
* Chronic steroid use
* Opioid use disorder
* Contraindication to performing any of the proposed blocks - active infection at the block site, systemic infection, allergy to local anesthetic medications
* Patients undergoing second surgery or urgent/emergent surgery
* Patients weighing < 50kg
* History of chronic pain and/or opioid tolerant
* Anticipated requirement for patient-controlled analgesia (PCA)
* Allergy or intolerance to any medication specified in the study protocol or postoperative pain management regimen
* Liver disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, PhD, MBA, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akerman M, Pejcic N, Velickovic I. A Review of the Quadratus Lumborum Block and ERAS. Front Med (Lausanne). 2018 Feb 26;5:44. doi: 10.3389/fmed.2018.00044. eCollection 2018. PMID 29536008
- [Background] Fang B, Wang Z, Huang X. Ultrasound-guided preoperative single-dose erector spinae plane block provides comparable analgesia to thoracic paravertebral block following thoracotomy: a single center randomized controlled double-blind study. Ann Transl Med. 2019 Apr;7(8):174. doi: 10.21037/atm.2019.03.53. PMID 31168455
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] MacFater WS, Rahiri JL, Lauti M, Su'a B, Hill AG. Intravenous lignocaine in colorectal surgery: a systematic review. ANZ J Surg. 2017 Nov;87(11):879-885. doi: 10.1111/ans.14084. Epub 2017 Jul 5. PMID 28677829
- [Background] Masic D, Liang E, Long C, Sterk EJ, Barbas B, Rech MA. Intravenous Lidocaine for Acute Pain: A Systematic Review. Pharmacotherapy. 2018 Dec;38(12):1250-1259. doi: 10.1002/phar.2189. Epub 2018 Nov 9. PMID 30303542
- [Background] Njathi CW, Johnson RL, Laughlin RS, Schroeder DR, Jacob AK, Kopp SL. Complications After Continuous Posterior Lumbar Plexus Blockade for Total Hip Arthroplasty: A Retrospective Cohort Study. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):446-450. doi: 10.1097/AAP.0000000000000589. PMID 28277419
- [Background] Shanthanna H, Moisuik P, O'Hare T, Srinathan S, Finley C, Paul J, Slinger P. Survey of Postoperative Regional Analgesia for Thoracoscopic Surgeries in Canada. J Cardiothorac Vasc Anesth. 2018 Aug;32(4):1750-1755. doi: 10.1053/j.jvca.2018.01.003. Epub 2018 Jan 5. PMID 29402627
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For 3 patients under the abdominal portion of this study, Erector Spinae Blocks were performed rather than Quadratus Lumborum Blocks. There are various anatomic reasons why a different block would be considered when performing the actual block. This study was analyzing Quadratus Lumborum Blocks for abdominal surgery, as such, the results from the patients who had Erector Spinae Blocks for abdominal surgery were excluded.
Groups:
- Continuous Nerve Blocks: A total of 7 subjects equally distributed to either continuous Erector Spinae Plane block for unilateral thoracic surgery, or continuous Quadratus Lumborum block for major abdominal surgery. Patients in this group will receive 20ml 0.5% ropivacaine per block performed after positioning of the needle followed by continuous perineural infusion of 0.25% lidocaine (10ml/hr) beginning in the post-anesthesia care unit (PACU) and continued for 72 hours or until 12 hours prior to patient discharge, whichever comes first, which is standard of care at this institution.
  Continuous Erector Spinae Plane Nerve Block: To be administered to subjects in the active comparator group receiving primary unilateral thoracic surgery.
  Continuous Quadratus Lumborum Nerve Block: To be administered to subjects in the active comparator group receiving primary major abdominal surgery.
  Ropivacaine 0.5% Injectable Solution: To be used in both treatment arms as nerve block initial bolus injection.
  Lidocaine: To be used perineurally as a 0.25% solution in the active comparator group at a rate of 10 ml/hr per perineural catheter.
- Single Nerve Blocks Plus IV Lidocaine Infusion: A total of 7 subjects equally distributed to either Erector Spinae Plane block for unilateral thoracic surgery, or Quadratus Lumborum block for major abdominal surgery, will be included . Patients in this group will receive 20ml 0.5% ropivacaine, 4mg dexamethasone, and 20mcg dexmedetomidine (30mcg if only one block is performed) per block after proper positioning of the Tuohy needle. Upon patient arrival in the recovery room a continuous infusion of IV lidocaine 50 mg /hr will be started and continued for 72 hours or until 12 hours prior to patient discharge, whichever comes first, which is standard of care at this institution.
  Single Erector Spinae Plane Nerve Block: To be administered to subjects in the experimental group receiving primary unilateral thoracic surgery.
  Single Quadratus Lumborum Nerve Block: To be administered to subjects in the experimental group receiving primary major abdominal surgery.
  Lidocaine IV: To be given postoperatively as a continuous infusion at a dose of 50 mg/hr in the experimental group.
  Ropivacaine 0.5% Injectable Solution: To be used in both treatment arms as nerve block initial bolus injection.
  Dexamethasone: To be used in the experimental arm as a nerve block adjuvant to promote prolonged single block duration, as is standard of care in this institution.
  Dexmedetomidine: To be used in the experimental arm as a nerve block adjuvant to promote prolonged single block duration, as is standard of care in this institution.
Period: Overall Study
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.86 (5.96) | 65.43 (7.72) | 68.64 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 78.29 (8.85) | 84.71 (14.90) | 81.50 (12.23)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption After Surgery
Description: Opioids will be converted to oral morphine equivalents
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: OME
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 7
OME | 34.93 (31.32) | 46.50 (33.37)

2. Secondary Outcome: Opioid Consumption After Surgery
Description: Opioids will be converted to oral morphine equivalents
Time Frame: 48 hours after surgery
Population: One patient from the single nerve block plus IV lidocaine infusion group was not included because they were discharged before 48 hours and opioids were not recorded as an outpatient.
Measure: Mean (Standard Deviation); unit: OME
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 6
OME | 61.5 (54.06) | 84.75 (65.57)

3. Secondary Outcome: Opioid Consumption After Surgery
Description: Opioids will be converted to oral morphine equivalents
Time Frame: 72 hours after surgery
Population: Two patients from the single nerve block plus IV lidocaine infusion group was not included because they were discharged before 72 hours and opioids were not recorded as an outpatient.
Measure: Mean (Standard Deviation); unit: OME
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 5
OME | 88.57 (60.24) | 128.1 (150.29)

4. Secondary Outcome: Pain After Surgery
Description: By numeric pain rating scale, 0 = no pain and 10 = worst possible pain
Time Frame: 6 hours after surgery
Population: One patient in the continuous nerve block group did not have pain scores recorded due to lethargy. They were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 6 | 7
score on a scale | 6.17 (3.25) | 6.14 (1.77)

5. Secondary Outcome: Pain After Surgery
Description: By numeric pain rating scale, 0 = no pain and 10 = worst possible pain
Time Frame: 12 hours after surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 6 | 7
score on a scale | 6.17 (3.67) | 6.07 (2.83)

6. Secondary Outcome: Pain After Surgery
Description: By numeric pain rating scale, 0 = no pain and 10 = worst possible pain
Time Frame: 24 hours after surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 6 | 7
score on a scale | 4.5 (2.17) | 6.43 (2.88)

7. Secondary Outcome: Pain After Surgery
Description: By numeric pain rating scale, 0 = no pain and 10 = worst possible pain
Time Frame: 48 hours after surgery
Population: One patient in the single nerve block plus IV lidocaine infusion group was discharged prior to 48 hours and did not have a pain score recorded at that time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 6
score on a scale | 5.86 (2.67) | 4.83 (3.37)

8. Secondary Outcome: Pain After Surgery
Description: By numeric pain rating scale, 0 = no pain and 10 = worst possible pain
Time Frame: 72 hours after surgery
Population: Three patients in the single nerve block plus IV lidocaine infusion group were discharged prior to 72 hours and did not have a pain score recorded at that time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 4
score on a scale | 5.36 (1.75) | 5.0 (1.83)

9. Secondary Outcome: Local Anesthetic Consumption After Surgery
Description: Local anesthetic consumption after surgery is reported in mg of lidocaine
Time Frame: 12 hours after surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 7
mg | 574.29 (179.73) | 600 (0)

10. Secondary Outcome: Local Anesthetic Consumption After Surgery
Description: Local anesthetic consumption after surgery is reported in mg of lidocaine
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 7
mg | 1096.07 (330.01) | 1139.29 (160.63)

11. Secondary Outcome: Local Anesthetic Consumption After Surgery
Description: Local anesthetic consumption after surgery is reported in mg of lidocaine
Time Frame: 48 hours after surgery
Population: One patient in the single nerve block plus IV lidocaine infusion group was discharged well before 48 hours, so their data was not included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 6
mg | 1973.57 (717.70) | 2308.33 (149.72)

12. Secondary Outcome: Local Anesthetic Consumption After Surgery
Description: Local anesthetic consumption after surgery is reported in mg of lidocaine
Time Frame: 72 hours after surgery
Population: Two patients in the single nerve block plus IV lidocaine infusion group were discharged well before 72 hours, so their data was not included.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 5
mg | 2721.79 (896.91) | 2570.0 (499.50)

13. Secondary Outcome: Serum Lidocaine Level
Description: Serum lidocaine level measured via a blood test. Lidocaine has a therapeutic drug range of 1.5 to 5.0 mcg/mL.
Time Frame: 24 hours after surgery
Population: Serum collection was not standard of care and was not collected for all participating subjects
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 2 | 0
mcg/mL | 2.5 (0) |

14. Secondary Outcome: Serum Lidocaine Level
Description: Serum lidocaine level measured via a blood test. Lidocaine has a therapeutic drug range of 1.5 to 5.0 mcg/mL.
Time Frame: 48 hours after surgery
Population: Serum collection was not standard of care and was not collected for all participating subjects
Measure: Number; unit: mcg/mL
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 0 | 1
mcg/mL |  | 5.8

15. Secondary Outcome: Serum Lidocaine Level
Description: Serum lidocaine level measured via a blood test. Lidocaine has a therapeutic drug range of 1.5 to 5.0 mcg/mL.
Time Frame: 72 hours after surgery
Population: Serum collection was not standard of care and was not collected for all participating subjects
Measure: Number; unit: mcg/mL
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 0 | 1
mcg/mL |  | 1.5

16. Secondary Outcome: Total Hospital Length of Stay
Description: Hospital length of stay is measured in days from admission until discharge.
Time Frame: From admission to discharge, on average 1-4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 7
days | 9.04 (6.50) | 4.94 (3.71)

17. Secondary Outcome: Incidence of Adverse Events
Description: Nausea and vomiting requiring treatment, hypotension, or bradycardia or tachycardia
Time Frame: From time of surgery to discharge, on average 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from hospital admission until hospital discharge. In this sample the timeline ranged from 1 day to 13 days.
Arm/Group | Continuous Nerve Blocks | Single Nerve Blocks Plus IV Lidocaine Infusion
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Nerve Blocks (N=7) | Single Nerve Blocks Plus IV Lidocaine Infusion (N=7)
Abnormal Lidocaine Blood Level (Product Issues) | 0 (0) | 1 (1) — Lidocaine levels reached 5.8mcg/mL which led to infusions being stopped. Normal lidocaine levels range between 1.5 and 5.0mcg/mL.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Nerve Blocks (N=7) | Single Nerve Blocks Plus IV Lidocaine Infusion (N=7)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) — Subject demonstrated abnormal lethargy; therefore, nerve blocks were paused for a day. Subject began antibiotics, showed signs of improvement, and peripheral nerve blocks were then restarted. Lethargy likely related to infection, not lidocaine.

LIMITATIONS AND CAVEATS:
We were not able to enroll enough subjects in a timely manner and our enrollment numbers did not reach the goal of our pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04208516/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04208516/ICF_001.pdf